CLINICAL TRIAL: NCT07242053
Title: Efficacy of Intraoperative CT Feedback of Wedge Resected Lung for the Assessment of Surgical Margin
Brief Title: Margin Intraoperative CT Feedback Feedback Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kazuhiro Yasufuku, Dr. Kazuhiro Yasufuku, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-5750
Record Dates: First submitted 2025-09-30; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: Surgical Margins
MeSH Terms: conditions — Lung Neoplasms; Disease; Margins of Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative CT of resected lung (Experimental)
  Interventions: Other: Intraoperative CT of resected lung

INTERVENTIONS:
Other: Intraoperative CT of resected lung — Once the wedge resection is performed, the resected specimen will brought for CT scan

SUMMARY:
To date, there is no established method for confirming whether sufficient margins have been obtained during surgery, only post-surgery by a pathologist. The purpose of this study is to evaluate the impact of intraoperative CT margin feedback on surgical decisions, such as additional removal. The ability to accurately evaluate surgical margins intraoperatively could reduce the risk of locoregional recurrence and eliminate the need for additional treatment after surgery. Moreover, optimal intraoperative feedback to surgeon could influence surgical decision making and contribute to the satisfactory outcome. This is a single center clinical trial. A total of 80 patients scheduled for wedge resections for lung malignancies (including suspected patients) will be enrolled in this study. Nine surgeons in the division of thoracic surgery will also be involved as participants. Once the wedge resection is performed, the resected specimen will be inflated and scanned by CT to measure surgical margin intraoperatively. Surgeons will have access to the CT data and the associated margin data immediately. They then may decide if an additional resection is required. The expected margin surveyed by questionnaire will be compared to CT measured margin, and CT measured margin will be compared to pathological margin questionnaires over course. After the total course of surgery, surgeons will be asked to complete a questionnaire as well to assess the satisfaction by intraoperative feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for wedge resection for lung malignancies (included suspected lesions).
* 18 years of age or older.

Exclusion Criteria:

* Any patients with inability to give informed consent
* Wedge resection for non-therapeutic purpose, e.g. diagnostic purpose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The contribution of intraoperative feedback to treatment decision, and its validity | 2 years
  After the total course of surgery, we will ask each surgeon individually for questionnaire 3 after feedback of the individual result of this study to assess the satisfaction by intraoperative feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT07242053/Prot_000.pdf